CLINICAL TRIAL: NCT01729078
Title: The Effects of Dietary Supplementation on Hepatic Insulin Action and Glucose Tolerance in Pre-diabetes
Brief Title: Dietary Interventions in Prediabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Rita Basu, PI, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 12-003216
Record Dates: First submitted 2012-11-09; First posted 2012-11-20 (Estimated); Last update posted 2015-07-29 (Estimated); Status verified 2015-07

CONDITIONS: Impaired Fasting Glucose; Pre Diabetes; Liver Fat
MeSH Terms: conditions — Glucose Intolerance; Fatty Liver | interventions — Diet Therapy

STUDY DESIGN:
Who Masked: Investigator

ARMS (3):
- high fat ( MUFA) diet (Experimental): intervention using high fat diet.
  Interventions: Dietary Supplement: Dietary intervention
- high carb/high fiber (Experimental): diet using high carb-high fiber with dry beans
  Interventions: Dietary Supplement: Dietary intervention
- high carb/low fat (Experimental): Habitual diet
  Interventions: Dietary Supplement: Dietary intervention

INTERVENTIONS:
Dietary Supplement: Dietary intervention — three different diets ( high fat-low carb-low fiber/high carb-low fat - high fiber/high carb-low fat-low fiber)

SUMMARY:
Assessment of glucose metabolism and liver fat after 12 week dietary intervention in pre diabetes subjects. Subjects will be randomized to either high fat (olive oil supplemented),high carb/high fiber (beans supplemented) and high carb/low fiber diets. Glucose metabolism will be assessed by labeled oral glucose tolerance test and liver fat by magnetic resonance spectroscopy pre randomization and at 8 and 12 week after starting dietary intervention.

ELIGIBILITY:
Inclusion Criteria:

* Impaired fasting glucose(100-125 mg/dl)
* HbA1c 5.7-6.4 %
* BMI 26-40 kg/sq.m

Exclusion Criteria:

* MRS contraindication
* Pregnant women
* Liver disease

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2012-10; Primary Completion 2013-10 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Changes in liver fat content after 12 weeks of intervention | 12 weeks

SECONDARY OUTCOMES:
Change in glucose metabolism after 12 weeks of intervention | 12 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Mayo clinic, Rochester, Minnesota, United States

REFERENCES:
- [Derived] Errazuriz I, Dube S, Slama M, Visentin R, Nayar S, O'Connor H, Cobelli C, Das SK, Basu A, Kremers WK, Port J, Basu R. Randomized Controlled Trial of a MUFA or Fiber-Rich Diet on Hepatic Fat in Prediabetes. J Clin Endocrinol Metab. 2017 May 1;102(5):1765-1774. doi: 10.1210/jc.2016-3722. PMID 28323952